CLINICAL TRIAL: NCT00844961
Title: Study of the Effectiveness of Internet Delivered Cognitive Behavior Therapy in a Sample of Consecutively Recruited Patients Diagnosed With Irritable Bowel Syndrome
Brief Title: Effectiveness of Internet Delivered Cognitive Behavior Therapy (CBT) for Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Allmänna arvsfonden (Unknown); Region Stockholm (Other Government); Königska-Söderströmska sjukhemmet (Unknown); Aleris Helse (Other)
Responsible Party: Nils Lindefors, Psykiatri Sydväst, Stockholms läns landsting
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-K
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2009-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; CBT; Internet treatment; Cognitive behavior therapy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet CBT (Experimental): 10 weeks of internet delivered cognitive behaviour therapy
  Interventions: Behavioral: Internet delivered cognitive behavior therapy
- Waiting list (No Intervention): Waiting list which is offered treatment after completion of post intervention assessments

INTERVENTIONS:
Behavioral: Internet delivered cognitive behavior therapy — 10 weeks of internet delivered cognitive behavior therapy targeted at reducing experience of IBS symptoms and improving quality of life. Patients are offered guidance via email by a therapist.
  Other Names: CBT
  Arms: Internet CBT

SUMMARY:
The study will recruit 80 out-patients diagnosed with Irritable Bowel Syndrome from a gastroenterological clinic. The recruitment will be consecutive with all patients receiving the diagnosis being offered to participate. After recruitment and 3 week baseline measure of IBS symptoms they will be randomised to either 10 weeks of internet delivered CBT or waiting list. After treatment IBS-symptoms are measured again to assess treatment effectiveness. All patients on waiting list are offered the same treatment as patients randomised to treatment.

All patients are assessed 12 months after completion of treatment.

Patients in treatment condition are hypothesized to experience significant reduction IBS symptoms and quality of life compared to patients on waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Irritable Bowel Syndrome according to Rome III criteria

Exclusion Criteria:

* History of inflammatory bowel disease (IBD)
* Symptom debut after age of 50
* Ongoing severe mental illness (psychosis, severe depression, suicidal ideation, bipolar disease)
* Inability to participate in internet delivered treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale - IBS Version (GSRS-IBS) | Before treatment
The Gastrointestinal Symptom Rating Scale - IBS Version (GSRS-IBS) | After treatment
The Gastrointestinal Symptom Rating Scale - IBS Version (GSRS-IBS) | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lindefors, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykatrienheten, M57, Psykiatri sydväst, Stockholm, Sweden

REFERENCES:
- [Derived] Ljotsson B, Andersson G, Andersson E, Hedman E, Lindfors P, Andreewitch S, Ruck C, Lindefors N. Acceptability, effectiveness, and cost-effectiveness of internet-based exposure treatment for irritable bowel syndrome in a clinical sample: a randomized controlled trial. BMC Gastroenterol. 2011 Oct 12;11:110. doi: 10.1186/1471-230X-11-110. PMID 21992655